CLINICAL TRIAL: NCT03400527
Title: The Effects of Self Directed Exercise on People With Fibromyalgia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shenandoah University (Other)
Responsible Party: Principal Investigator, AJ Lievre, Assistant Professor, Shenandoah University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SUPT 5
Record Dates: First submitted 2018-01-08; First posted 2018-01-17 (Actual); Last update posted 2018-04-24 (Actual); Status verified 2018-04

CONDITIONS: Fibromyalgia
MeSH Terms: conditions — Fibromyalgia | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Exercise (Experimental): Participant will be pedaling a stationary exercise bicycle
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Exercise — Participants will pedal on a stationary bicycle up to 25 minutes 2-3 times a week for 4 weeks at a self directed pace and intensity

SUMMARY:
The purpose of this study is to determine the effects of self directed exercise on pain and function reported in patients with Fibromyalgia both in the short term and long term. Previous studies have shown that patients with fibromyalgia respond better to a single session of self directed exercise compared to prescriptive exercise. To the investigator's knowledge, no studies have examined the impact on pain and function after multiple sessions of self directed exercise in this patient population.

This study hoes to be a case series exploring the effects of self directed exercise on participants with fibromyalgia. Participants will be encouraged to exercise 8-12 times in a 4 week time frame at a self selected pace and intensity on a stationary bicycle. Outcome measures such as the Fibromyalgia Impact Questionnaire, SF-36 and Numeric Pain Rating Scale will be used prior to study participation as well as 4 and 8 weeks following the start of participation.

ELIGIBILITY:
Inclusion Criteria:

* over the age of 18
* a medical diagnosis of Fibromyalgia
* sedentary level of activity prior to entry. Sedentary level of activity is defined as: no participation in regular physical activity more strenuous than slow paced walking for a maximum of 2 times per week for the 4 months prior to study entry.
* signed release from their physician stating that they are able to participate in the study.

Exclusion Criteria:

* presence of an acute or chronic medical condition such as cancer
* infection, cardiovascular or respiratory disease (that would limit their exercise participation), metabolic or musculoskeletal or neurologic condition (systemic lupus or rheumatoid arthritis, or other pain disorders)
* already participating or plan on participating in a regular aerobic exercise program 6 months prior to the study
* ongoing or planned Physical Therapy treatment
* drug dependency

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2018-03-30 (Actual); Primary Completion 2018-09 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Change in Fibromyalgia Impact Questionnaire | 0, 4 and 8 weeks
  An instrument developed to assess the current health status of women with the fibromyalgia syndrome in clinical and research settings1.
  Assesses current health and functional status in people with Fibromyalgia

SECONDARY OUTCOMES:
Change in Numeric Pain Rating Scale | 0, 4 and 8 weeks
  Paint rating scale from 0-10
Change in Short Form (SF) - 36 | 0, 4 and 8 weeks
  Survey of reported health

CONTACTS AND LOCATIONS:
Locations (1):
- Woodstock Rehab & Fitness, Woodstock, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ellingson LD, Stegner AJ, Schwabacher IJ, Koltyn KF, Cook DB. Exercise Strengthens Central Nervous System Modulation of Pain in Fibromyalgia. Brain Sci. 2016 Feb 26;6(1):8. doi: 10.3390/brainsci6010008. PMID 26927193